CLINICAL TRIAL: NCT02166138
Title: Non-Ablative Fractional Resurfacing of Total Knee Replacement Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles Cornell, MD (Other)
Responsible Party: Sponsor-Investigator, Charles Cornell, MD, MD, Hospital for Special Surgery, New York
Organization: Hospital for Special Surgery, New York (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13045
Record Dates: First submitted 2014-05-31; First posted 2014-06-18 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Epidermal Thickening, Unspecified

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Laser treated Group (Experimental): Patients in this group will be given the laser treatment with the non-abilative 1540 nm wavelength. Patients will be blinded to this procedure as they will be wearing protective eye wear and noise canceling headphones. These patients will undergo the treatment 3 times, one at day of discharge, second at the 4 week follow up visit, and third at the 8 week follow up visit. After the 8 week follow up visit, patients will be asked to come in for the 3 month follow up visit and 1 year follow up visit for an evaluation. At each visit, the patient's scar will be photograph for evaluation. Each patient will also be asked to fill out the POSAS, and KOOS at each follow up visits. Thus, patients in this group will be getting the Non-Abilative laser treatment.
  Interventions: Procedure: Non-Abilative Laser treatment
- Not Laser treated Group (Placebo Comparator): Patients in this group will be given the laser treatment with the 1540 non-abilative laser device, but the device will not be set to provide treatment. Patients will be blinded to this procedure as they will be wearing protective eye wear and noise canceling headphones. These patients will undergo the treatment 3 times, one at day of discharge, second at the 4 week follow up visit, and third at the 8 week follow up visit. After the 8 week follow up visit, patients will be asked to come in for the 3 month follow up visit and 1 year follow up visit for an evaluation. At each visit, the patient's scar will be photograph for evaluation. Each patient will also be asked to fill out the POSAS, and KOOS at each follow up visits.

INTERVENTIONS:
Procedure: Non-Abilative Laser treatment — Patients in this group will be given the laser treatment with the non-abilative 1540 nm wavelength. Patients will be blinded to this procedure as they will be wearing protective eye wear and noise canceling headphones. These patients will undergo the treatment 3 times, one at day of discharge, second at the 4 week follow up visit, and third at the 8 week follow up visit. After the 8 week follow up visit, patients will be asked to come in for the 3 month follow up visit and 1 year follow up visit for an evaluation. At each visit, the patient's scar will be photograph for evaluation. Each patient will also be asked to fill out the POSAS, and KOOS at each follow up visits.
  Other Names: Laser treated group
  Arms: Laser treated Group

SUMMARY:
The condition to be studied is post-surgical scarring following primary total knee replacement, specifically whether fractional non-ablative laser therapy can be used to significantly decrease the morbidity of scarring.

DETAILED DESCRIPTION:
Patients undergoing unilateral, primary total knee replacement will be enrolled in the study in the treating surgeon's office at the time surgery is indicated and scheduled. Patient's will be asked to enroll in the study if they are indicated by the treating surgeon for primary total knee replacement, are 18 years of age or older, and, if they have no history of wound healing problems, chronic infection or connective tissue disorder and if they have a Fitzpatrick skin type between I and VI. Patients will be excluded from the study if they: have any prior history of surgery on the indicated knee; have a mental or psychological illness that prohibits them from consenting or completing the necessary forms; if they refuse to consent to be in the study; or, if they have a history of wound healing problems, or a diagnosed skin or connective tissue disease. Standard baseline health information and demographics will be collected at the time of enrollment (gender, age, co-morbidities, etc.).

On the day of surgery, patients will be randomized to have their surgical incision treated with the non-ablative fractional laser or treated with the placebo laser. Randomization will be computer-generated and stored in opaque sealed envelopes. For each patient, randomization will take place prior to surgery in the holding area on the day of surgery. At discharge, the laser technician will open the sealed envelope to reveal the allocation into control or experimental groups. The technician will then treat the patient appropriately as per the protocol. Proper randomization will be ensured by the technician, principal investigator and co-investigators. The patients, principal investigator and co-investigators collecting the data will be blinded to the randomization. The technician providing the laser therapy will not be blinded.

The incisional length will be determined by the treating surgeon at the time of surgery based on what he deems will be adequate given the patient's body habitus and the technical demands of the surgery. The skin incision will always be made with a new, sharp, sterile 10 blade. Subcutaneous dissection will be done with the scalpel as well.

Closure of the wound will be done with 0-vicryl sutures for the arthrotomy and deep subcutaneous tissue. The sutures will be tied in an interrupted simple pattern. The superficial subcutaneous tissue layer will be closed with interrupted buried 2.0-vicryl sutures. The skin will be closed with a 4.0 monocryl running subcuticular stitch. The wound will be dressed with a sterile dressing that will come off on post operative day two.

After the primary dressing is taken down, the wound will be left open to air unless there is active drainage. If active drainage is present, sterile gauze will be kept on the wound until it is dry.

As a dry wound is a pre-requisite for patient discharge, no patient will be discharged with a draining wound. On the day of discharge, the patient will have the first of the non-ablative, fractional laser treatments done in the hospital. This will be performed by a registered technician who has been trained in the use of the non-ablative, fractional laser. The technician will be trained by the company providing the device and will have completed the hospital's required laser training prior to using the device on patients.

The laser settings will be preset at 15 mjs and 50 mj. The number of passes used per patients will be 5 passes, and this is determined by the plastic surgeon included on the study and will be individualized to the patient's Fitzpatrick skin type. The technician will know the status of the patient's randomization and will either treat the patient with the laser or turn the laser on and apply it in the standard fashion without activating the device. The technician will also apply a Lidocaine patch in order to numb the area that will be treated by the laser device and keep the patient blinded from the treatment. The patients will be asked to wear opaque glasses that prevent them from seeing the technician using the laser so as to remain blinded to the treatment. Additionally, they will be asked to wear noise-cancelling headphones so as to minimize any sound the active laser makes.

On the day of discharge the patient will have the first of the non-ablative, fractional laser treatments performed in the hospital by the registered technician who has been trained in the use of the non-ablative fractional laser. The patients will be given strict instruction in a standardized wound care regimen. They will complete a standard post TKR rehabilitative course. At the 4-week and 8-week time points the patient will return to the clinic for a wound check and for the 2nd and 3rd laser therapy treatment. The patients will see the surgeon at the 4-week follow up visit, as this is standard of care. At week 8,the non-Standard of Care visit, the treating surgeon's nurse and the laser technician will see the patients. If the patient, nurse or technician has any concerns about the status of the wound, the Principle Investigator will be notified. Patients will not be charged for the 8-week visit.

At the 4 week, 8 week, 3 month and 1 year visits the surgical scar will be photographed in a standardized, controlled fashion. Dr. Rothaus, a plastic surgeon, has extensive experience with standardized cosmetic photography and will provide his expertise. Briefly, the same camera, lens, lighting and position will be used for all patients at all time points. The goal is to have the only variable be the appearance of the scar. At each of these visits, the patient will complete a validated scar assessment outcomes tool, the Patient and Observer Scar Assessment Scale (POSAS).(22) Additionally, one of three experts (Dr. Rothaus, Ms. Trezza, Dr. Cornell) trained in scar assessment will inspect the patient's scar and complete the observer portion of the scar assessment instrument. In addition to the POSAS, each patient will also complete a valid knee outcomes instrument, the Knee Injury and Osteoarthritis Outcome Score (KOOS)(23) at each visit. The data will be collected in the physician's private office prior to the scheduled surgery and after surgery at each visit. An identified co-investigator, with the appropriate HIPAA and human subjects research training will be responsible for administering the knee instruments, answering any of the patient's questions, and then collecting the instruments after they have been completed. This will ensure that the surgeon does not have access to the patient's responses.

The primary outcome will be the difference in POSAS score between patients treated with the laser and those treated with placebo. Secondary outcomes include the difference in POSAS observer score as well as the difference in KOOS score between the experimental and the control group.

While the investigators group is the first to use this technology on Total Knee Replacement scars, Vasily et al. in 2009 reported on the effectiveness of laser treatment of post-surgical and traumatic scars and found that relative to baseline, 73% of scars improved 50%, and 43% improved by 75% or more. Overall, all of the treated scars demonstrated some clinical improvement with a mean overall improvement of 52%. Side effects were minimal and included swelling (95%), erythema (94%) and purpura (5%).(9) All side effects completely resolved at the one-month follow-up visit.

Additionaly, the investigators pilot study has demonstrated that the laser treatment is safe, as the investigators have applied the treatments to ten patients, in the manor mentioned above, and have not seen any complications thus far. On the basis of this data and the pilot study, treatment with the non-ablative fractional laser has been deemed both safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if:

  * They are indicated for primary total knee replacement
  * Have no history of wound healing problems, chronic infection, or known skin or connective tissue disease.
  * Are 18 years of age or older
  * Have a skin type classified as a Fitzpatrick type I-VI.

Exclusion Criteria:

* Patients will be excluded for the following reasons:

  * Any prior history of surgery on their knee
  * Mental or psychological illness that prohibits the patient from completing the necessary forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
The change in POSAS scores between patients in the laser treated group and the not laser treated group at 4 weeks, 8 weeks, 3 month, and 1 year follow up visits. | 4 week, 8 week, 3 month, and 1 year follow up visits
  The primary outcome will be the difference in patient reported POSAS score between those patients that received laser therapy and those who did not receive laser therapy. The POSAS will be collected at the 4 week, 8 week, 3 month and 12 month time points.
  The POSAS consists of two scales: the patient scale and the observer scale. Both scales consist of six items that are scored numerically. The six items on the observer scale are: scar vascularity, pigmentation, pliability, thickness, relief and surface area. The six items scored by patients are: pain, itching, color, pliability, thickness and relief. Each of the six items is scored from 1-10 with 10 indicating the worst imaginable scar outcome. Each of the scores for the six items is added up for a cumulative score between 6 and 60 where 6 represents normal skin and 60 represents the worst scar imaginable. Both the patient and observer scale have been found to be reliable and valid in the evaluation of linear, surgical scars.

SECONDARY OUTCOMES:
KOOS | 4 week, 8 week, 3 month, and 1 year follow up visits
  Secondary outcomes include the difference in Knee injury and Osteoarthritis Outcome Score KOOS score at 4 week, 8 week, 3 months and 1 year between the treated and untreated groups. Additionally, any data collected at routine follow-ups will be collected and analyzed. This includes baseline demographic information as well as physical exam findings, including pre-operative and post-operative knee range of motion (ROM).
  The KOOS adopted the Western Ontario and McMaster Universities Arthritis Index and added two additional subscales to evaluate knee function after ligament, articular cartilage, or meniscal injury, and their respective treatments. The KOOS proved to be a patient-oriented outcome measure and demonstrated test-retest reliability and internal consistency. It was found to be more responsive than the WOMAC and SF-36, and validation was performed for face, content, criterion, concurrent, construct and convergent validity.

CONTACTS AND LOCATIONS:
Overall Officials: Charles N. Cornell, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Lupton JR, Alster TS. Laser scar revision. Dermatol Clin. 2002 Jan;20(1):55-65. doi: 10.1016/s0733-8635(03)00045-7. PMID 11859594
- [Background] Atkinson JA, McKenna KT, Barnett AG, McGrath DJ, Rudd M. A randomized, controlled trial to determine the efficacy of paper tape in preventing hypertrophic scar formation in surgical incisions that traverse Langer's skin tension lines. Plast Reconstr Surg. 2005 Nov;116(6):1648-56; discussion 1657-8. doi: 10.1097/01.prs.0000187147.73963.a5. PMID 16267427
- [Background] Baisch A, Riedel F. [Hyperplastic scars and keloids. Part I: basics and prevention]. HNO. 2006 Nov;54(11):893-904; quiz 905. doi: 10.1007/s00106-006-1462-z. German. PMID 17041777
- [Background] O'Brien L, Pandit A. Silicon gel sheeting for preventing and treating hypertrophic and keloid scars. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD003826. doi: 10.1002/14651858.CD003826.pub2. PMID 16437463
- [Background] Bock O, Schmid-Ott G, Malewski P, Mrowietz U. Quality of life of patients with keloid and hypertrophic scarring. Arch Dermatol Res. 2006 Apr;297(10):433-8. doi: 10.1007/s00403-006-0651-7. Epub 2006 Mar 10. PMID 16528552
- [Background] Khanna A, Gougoulias N, Longo UG, Maffulli N. Minimally invasive total knee arthroplasty: a systematic review. Orthop Clin North Am. 2009 Oct;40(4):479-89, viii. doi: 10.1016/j.ocl.2009.05.003. PMID 19773053
- [Background] Mow CS, Woolson ST, Ngarmukos SG, Park EH, Lorenz HP. Comparison of scars from total hip replacements done with a standard or a mini-incision. Clin Orthop Relat Res. 2005 Dec;441:80-5. doi: 10.1097/01.blo.0000191317.85422.c3. PMID 16330988
- [Background] Tanzi EL, Lupton JR, Alster TS. Lasers in dermatology: four decades of progress. J Am Acad Dermatol. 2003 Jul;49(1):1-31; quiz 31-4. doi: 10.1067/mjd.2003.582. PMID 12833005
- [Background] Vasily DB, Cerino ME, Ziselman EM, Zeina ST. Non-ablative fractional resurfacing of surgical and post-traumatic scars. J Drugs Dermatol. 2009 Nov;8(11):998-1005. PMID 19894367
- [Background] Haedersdal M, Moreau KE, Beyer DM, Nymann P, Alsbjorn B. Fractional nonablative 1540 nm laser resurfacing for thermal burn scars: a randomized controlled trial. Lasers Surg Med. 2009 Mar;41(3):189-95. doi: 10.1002/lsm.20756. PMID 19291747
- [Background] Hedelund L, Moreau KE, Beyer DM, Nymann P, Haedersdal M. Fractional nonablative 1,540-nm laser resurfacing of atrophic acne scars. A randomized controlled trial with blinded response evaluation. Lasers Med Sci. 2010 Sep;25(5):749-54. doi: 10.1007/s10103-010-0801-1. Epub 2010 Jun 17. PMID 20556471
- [Background] Laubach HJ, Tannous Z, Anderson RR, Manstein D. Skin responses to fractional photothermolysis. Lasers Surg Med. 2006 Feb;38(2):142-9. doi: 10.1002/lsm.20254. PMID 16392146
- [Background] Orringer JS, Rittie L, Baker D, Voorhees JJ, Fisher G. Molecular mechanisms of nonablative fractionated laser resurfacing. Br J Dermatol. 2010 Oct;163(4):757-68. doi: 10.1111/j.1365-2133.2010.09998.x. PMID 20854401
- [Background] Sherling M, Friedman PM, Adrian R, Burns AJ, Conn H, Fitzpatrick R, Gregory R, Kilmer S, Lask G, Narurkar V, Katz TM, Avram M. Consensus recommendations on the use of an erbium-doped 1,550-nm fractionated laser and its applications in dermatologic laser surgery. Dermatol Surg. 2010 Apr;36(4):461-9. doi: 10.1111/j.1524-4725.2010.01483.x. Epub 2010 Feb 19. PMID 20187898
- [Background] Badawi A, Tome MA, Atteya A, Sami N, Morsy IA. Retrospective analysis of non-ablative scar treatment in dark skin types using the sub-millisecond Nd:YAG 1,064 nm laser. Lasers Surg Med. 2011 Feb;43(2):130-6. doi: 10.1002/lsm.21031. PMID 21384394
- [Background] Fitzpatrick TB. Soleil et peau. J Med Esthet 1975;2:33-4.
- [Background] Carvalho RL, Alcantara PS, Kamamoto F, Cressoni MD, Casarotto RA. Effects of low-level laser therapy on pain and scar formation after inguinal herniation surgery: a randomized controlled single-blind study. Photomed Laser Surg. 2010 Jun;28(3):417-22. doi: 10.1089/pho.2009.2548. PMID 19821701
- [Background] Conologue TD, Norwood C. Treatment of surgical scars with the cryogen-cooled 595 nm pulsed dye laser starting on the day of suture removal. Dermatol Surg. 2006 Jan;32(1):13-20. doi: 10.1111/1524-4725.2006.32002. PMID 16393593
- [Background] Kim SG, Kim EY, Kim YJ, Lee SI. The Efficacy and Safety of Ablative Fractional Resurfacing Using a 2,940-Nm Er:YAG Laser for Traumatic Scars in the Early Posttraumatic Period. Arch Plast Surg. 2012 May;39(3):232-7. doi: 10.5999/aps.2012.39.3.232. Epub 2012 May 10. PMID 22783532
- [Background] Nouri K, Jimenez GP, Harrison-Balestra C, Elgart GW. 585-nm pulsed dye laser in the treatment of surgical scars starting on the suture removal day. Dermatol Surg. 2003 Jan;29(1):65-73; discussion 73. doi: 10.1046/j.1524-4725.2003.29014.x. PMID 12534515
- [Background] Pham AM, Greene RM, Woolery-Lloyd H, Kaufman J, Grunebaum LD. 1550-nm nonablative laser resurfacing for facial surgical scars. Arch Facial Plast Surg. 2011 May-Jun;13(3):203-10. doi: 10.1001/archfacial.2011.28. PMID 21576668
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417